CLINICAL TRIAL: NCT02302885
Title: Human Blood Collection to Serve as Negative Control for Validation of Circulating Tumor Cell Assay
Brief Title: Healthy Human Control Blood Collection for Validation of Biomarker Assay
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 42914
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: cancer-free 18-60 year old men and women
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — About 20 mL blood will be collected from volunteers up to 20 different timepoints.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood collection — Blood Collection

SUMMARY:
Human blood will be collected to serve as control in validating clinical studies studying the detection and levels of circulating tumor cells and microvesicles in cancer patients. Targeted population is cancer-free 18-60 year old men and women. Volunteer selection will rely upon a short health questionnaire. About 20 mL blood will be collected from volunteers up to 20 different timepoints. The Procedure involves minimal risk of harm (eg discomfort, bruising) to the volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-60 years old Gender: Male and Female

Exclusion Criteria:

* No previously diagnosed malignancy Age: It is important to obtain a healthy, cancer-free volunteer population to serve as negative controls for this detection assay.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: cancer-free 18-60 year old men and women
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
blood count | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jay Dorsey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States